CLINICAL TRIAL: NCT06396650
Title: Assessment of Fall Risks and Subject-specific Training for Fall Reduction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Li-Qun Zhang, Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HP-00108616-
Record Dates: First submitted 2024-04-22; First posted 2024-05-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Fall Risk
Keywords: Fall prevention; Perturbation training; Multidirectional perturbation; Home-based training; Subject-specific training strategy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lab and home-based training (Experimental): Conduct balance training and/or lower-limb muscle strengthening in lab and at home
  Interventions: Device: Home-based training; Device: Lab-based training

INTERVENTIONS:
Device: Home-based training — 1. If the participant shows instability in any specific perturbation directions or with excessive body swaying, the participant will practice walking with a cellphone strapped on the chest in-home training. A cellphone App will detect potential excessive body swaying in any directions and prompt the participant with real time audio-visual feedback to reduce sway in the specific directions.
  2. If the subject is diagnosed with collapse-related vertical instability, lower-limb muscle strengthening will be emphasized in the training. The subject may work out with a Shuttle Mini-Press, AB Squat machine, Rowing machine, or Upright Row-n-Ride. The Investigators will select one machine appropriate for the subject to take home. The exercise will be 3-5 sets a day and about 15 repetitions per set. In the beginning, the exercise can be slower and with fewer repetitions based on the subject's capability. As the subject progresses, the subject may change from one exercise machine to another.
Device: Lab-based training — In the weekly lab-based training session, the subject will do individualized training using the sliding stepping trainer, with a focus on the direction the subject showed higher risks of falling, as identified in the initial assessment. The sliding stepping trainer will generate perturbations of the footplates in those identified risky directions during stepping.

SUMMARY:
The target population of this project is older people with high risks of falls. About 30% community-dwelling individuals over 65 years of age fall each year and the rate of fall related injuries leading to loss of function and independence increases with age. Falls are the leading cause of fatal and non-fatal injuries and the leading cause traumatic brain injury in older adults. Slip-related falls in older adults comprise 40% of outdoor falls and are the leading cause of hip fracture or traumatic head injury. In 2012, 2.4 million non-fatal falls were treated in emergency room visits with $30 billion dollars spent on direct medical costs. In addition to fractures and traumatic brain injury, nonfatal falls frequently lead to reduced levels of activity, fear of falling, and reduced quality of life. Clearly, advancing the predictive, preventative, and rehabilitative methods aimed at reducing the risk of injurious falls in this population is imperative. Although falls are multi-factorial in nature, there has been few individualized assessment of the biomechanical causes of falls.

The purpose of this study is to conduct subject-specific training on older adults with fall risks with combined home-hospital rehabilitation. This project will involve rehabilitation interventions based on the characteristics of falling patterns and older adults with reduced capability controlling the balance. To conduct subject-specific fall prevention training. based on identified individual fall mechanisms.

DETAILED DESCRIPTION:
Forty older adults (study group) with high risk of fall (i.e. with one or more fall in the past 12 months) will be recruited. The fall mechanisms will be examined in previous Aims 1 and 2 part of this study.

Assessments will be conducted to identify the fall risks and falling mechanisms by measuring subjects' responses to the movements of the footplates the subject stands on. Training procedures will then be designed for each subject, including training both in the research lab (once per week) and at home (three times per week) for six weeks. The subject will also revisit the lab for a follow-up assessment two months after the 6-week training.

Based on the identified falling mechanisms, a specific training for each subject will be set up using the sliding stepping fall rehabilitation system for one session per week over six weeks in the lab. The participants will also do home training exercises 3 times per week after initial in-lab instructed training. Participants will come to the lab and have biomechanical and clinical evaluations before and after the 6-week training (called Pre & Post), and then at a two-month follow-up as the final evaluation for total three times of evaluations.

All the subjects will be informed about the experimental procedures, and sign an IRB approved consent form prior to study participation and experimental tests.

All participants will be protected from the risk of falling with a harness system. The harness is mounted in mobile cart. A researcher will push the mobile cart following the participant's walking while walking on the ground.

Home-based training: The older adults will also undergo corresponding home-based training. Training at home may include normal walking and strength training based on the results in-lab assessments for each older adult and research team instructions.

1. . If the participant shows instability during walking in any specific perturbation directions or with excessive body swaying (left-right, forward-backward, or any oblique directions) based on the initial lab assessment, the participant will practice walking with a cellphone strapped on the chest in home training. A cellphone App will detect potential excessive body swaying in any directions and prompt the participant with real time audio-visual feedback to reduce sway in the specific directions. During the walking training at home, the participant will set up for a distance of a few meters to walk and repeat the walking distance for 12 to 15 times in a slow speed. the participant can take short break between the walking trials.

   1. For protection of falling risk, the participant needs to have a family member to help check the walking ground first before the walking to make sure the ground condition is good and clean.
   2. If the participant uses a cane or walker regularly, the participant will continue using the cane or walker during training at home with the cellphone attached.
   3. The participant should be monitored by a family member while doing the training at home.
   4. Training improvement will be evaluated in the weekly lab session. It is possible to make adjustment of the training program as the participant progresses.
2. . If the subject is diagnosed with collapse-related vertical instability associated with falls, lower-limb muscle strengthening will be emphasized in the training. The subject may work out with a Shuttle Mini-Press, AB Squat machine, Rowing machine, or Upright Row-n-Ride at home. The several exercise machines are similar to each other in strengthening the lower limb muscles but the challenging level gradually increasing. The Shuttle Mini Press allows the subject to train in stable seated or in-bed postures. The AB Squat machine allows squatting exercise with the two feet always on the ground. The rower allows seated sliding training. The Upright Row-n-Ride allows training in up-and-down fashion. The research team will select one machine appropriate for the subject to take home. The exercise will be 3-5 sets a day and about 15 repetitions per set. In the beginning, the exercise can be slower and with fewer repetitions based on the subject's capability. The subject can take a short break between the strength training sets. As the subject progresses, the subject may change from one exercise machine to another.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 to 85 years old
2. Have a family member at home for safety.
3. There is no severe injury or pain at the lower extremities.
4. With one or more falls in the past 12 months or walk with instability
5. Individuals who are taking medication, there should be no planned medication changes for the study duration of 3.5 months.
6. All the participants should be capable of independent walking.

Exclusion Criteria:

1. Enrollment in another lower limb rehabilitation program;
2. severe pain in the lower limbs;
3. previous myocardial infarction
4. Body weight over 280 lbs
5. Cognitive impairment (Mini-Mental Status Examination (MMSE) score less than 25)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Fall risks | The first visit, immediately after the training, and a follow-up evaluation session two-month after the training
  Berg Balance Scale (BBS) evaluation will be used which provides a value for fall risks assessment.

SECONDARY OUTCOMES:
Lower limb muscle strength | The first visit, immediately after the training, and a follow-up evaluation session two-month after the training
  The lower limb muscle strength will be measured manually by a researcher using dynamometry
Ground impact forces captured by forces plates during walking | The first visit, immediately after the training, and a follow-up evaluation session two-month after the training
  Subjects' ground impact forces captured by forces plates during multidirectional perturbations during walking.
Body kinematcis during walking | The first visit, immediately after the training, and a follow-up evaluation session two-month after the training
  Subjects' body kinematics measured by wearable IMUs during multidirectional perturbations during walking.
Body reactions against perturbations | The first visit, immediately after the training, and a follow-up evaluation session two-month after the training
  Subjects' body reactions to multidirectional perturbations during walking. Reactions include loss of balance, recovery steps, and falls, which will be identified by videos.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Qun Zhang, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Baltimore, Baltimore, Maryland, United States